CLINICAL TRIAL: NCT03462017
Title: Study to Assess the Pharmacodynamic Effects of Repeated Oral Doses of SAR247799 on Endothelial Function in Male and Female Patients With Type 2 Diabetes Mellitus
Brief Title: Pharmacodynamic Study to Assess the Effects of Repeated Dosing of SAR247799 on Endothelial Function in Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Basic Science
Other Study IDs: PDY15286; 2017-002592-26 (EudraCT Number); U1111-1197-8124 (Other: UTN)
Record Dates: First submitted 2018-03-06; First posted 2018-03-12 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Microvascular Coronary Artery Disease
MeSH Terms: interventions — Sildenafil Citrate; Acetylcholine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- SAR247799 (Experimental): SAR247799 repeated doses once daily in the morning under fasted condition for 28 days according to a sequential dose design
  Interventions: Drug: SAR247799; Drug: Acetylcholine
- Placebo (Placebo Comparator): Identical matching placebo for SAR247799 and for sildenafil once daily in the morning under fasted condition for 28 days
  Interventions: Drug: Placebo; Drug: Acetylcholine
- Sildenafil (Active Comparator): Sildenafil once daily in the morning under fasted condition for 28 days
  Interventions: Drug: Sildenafil; Drug: Acetylcholine

INTERVENTIONS:
Drug: SAR247799 — Pharmaceutical form:Capsule Route of administration: Oral
  Arms: SAR247799
Drug: Placebo — Pharmaceutical form:Capsule Route of administration: Oral
  Arms: Placebo
Drug: Sildenafil — Pharmaceutical form:Encapsulated tablet Route of administration: Oral
  Arms: Sildenafil
Drug: Acetylcholine — Pharmaceutical form:Solution Route of administration: Transdermal

SUMMARY:
Primary Objective:

To assess the pharmacodynamic effects of SAR247799 on macrovascular endothelial function of the brachial artery using flow-mediated dilation (FMD) in patients with type 2 diabetes mellitus (T2DM).

Secondary Objective:

* To assess the pharmacodynamic effects of SAR247799 on microvascular endothelial function using laser Doppler perfusion monitoring in patients with T2DM.
* To assess the safety profile of SAR247799 in patients with T2DM.
* To assess the plasma pharmacokinetic profile of SAR247799 in patients with T2DM.

DETAILED DESCRIPTION:
Study duration per patient is approximately 10 weeks including a 4-week treatment period.

ELIGIBILITY:
Inclusion criteria :

* Male and female stable Type 2 diabetes mellitus (T2DM) patients.
* Body Mass Index between 18 and 35 kg/m^2.
* Stable T2DM patients, but otherwise healthy as assessed by a clinical and laboratory assessments and detailed medical history.
* Diagnosis of T2DM for at least 6 months at the time of the screening visit.
* Glycosylated hemoglobin (HbA1c) < 8.5%.
* estimated glomerular filtration rate ˃60 mL/min/1.73 m^2.
* Flow-mediated dilatation (FMD) ≤7% at screening.
* Treatment of T2DM with lifestyle interventions or stable oral antidiabetic treatment for at least 3 months prior to inclusion.
* No clinically significant abnormality detected in cardiac echography, as assessed by certified Cardiologist, performed at screening.

Exclusion criteria:

* Any history or presence of clinically relevant or symptomatic gastrointestinal, hepatic, metabolic (except stable T2DM and controlled dyslipidemia), hematological, osteomuscular, articular, psychiatric, systemic, gynecologic (if female), or infectious disease, or ongoing cancer (including basal cell skin carcinoma), or signs of acute illness which as judged by the Investigator, may affect the patient's participation in or the outcome of this study.
* Symptomatic postural hypotension, irrespective of the decrease in blood pressure, or asymptomatic postural hypotension defined as a decrease in systolic blood pressure ≥30 mmHg within 3 minutes when changing from 10 min supine to standing position, at screening.
* History of symptomatic bradycardia, fainting, collapse, syncope, or vasovagal reactions in the last 6 months.
* Presence or history of drug hypersensitivity and/or allergy to any ingredients of the investigational product and/or non-investigational product diagnosed and treated by a physician.
* Any subject who cannot be treated with sildenafil because of conditions mentioned in the contra-indication, warning and precautions sections of sildenafil product information notably subjects with anatomical deformity of the penis.
* Loss of vision due to non-arteritic, neuro-optic, anterior ischemia assessed in ophtalmologic examination at screening.
* If female, pregnancy (defined as positive β-human chorionic gonadotropin blood and urine test), breast-feeding.
* Generally any medication which has a potential to interfere with the safety, pharmacokinetics of SAR247799 and sildenafil, or with study measurements is not allowed, and in particular:
* Nitrates, all calcium channel blockers, phosphodiesterase type 5 inhibitors (except investigational medicinal product [IMP]), guanylate cyclase stimulators use or anticipated during the study;
* Beta-blockers;
* Glucagon-like peptide-1 agonists;
* Insulins (all types);
* Anticoagulants, antithrombotics except aspirin;
* Any drugs which decrease heart rate;
* Antiarrhythmics;
* Digoxin;
* Cholinergic agents eg pilocarpine or cholinesterase inhibitors eg neostigmine, guanidine;
* Recent (≤3 months) use of systemic immunosuppressive or corticosteroid therapy;
* Any inactivated vaccination (eg, seasonal influenza) during study treatment, any attenuated vaccination within 2 months before inclusion, and any biologics (antibody or its derivatives) given within 4 months before inclusion;
* Any consumption of citrus fruits (grapefruit, orange, etc) or their juices within 3 days before inclusion as weak inhibitor of CYP3A4 gut wall metabolism.
* Any severe dyslipidemia with fasting triglycerides > 450 mg/dL.
* Any hyperosmolar hyperglycemic episode with severe neurological symptoms (eg, coma, aphasia) in the last 3 months before screening.
* Weight change of ≥5 kg during the last 2 months prior to screening.
* History or presence of clinically relevant or symptomatic pulmonary disease, such as asthma, chronic obstructive pulmonary disease, pulmonary embolism, pulmonary fibrosis, pulmonary hypertension which as judged by the Investigator, may affect the patient's participation in or the outcome of this study.
* Cardiovascular history such as:
* History or presence of a clinically relevant or symptomatic cardiovascular disease such as acute coronary syndrome (ACS), stroke, transient ischemic accident (TIA), obstructive or congestive heart failure, or structural heart disease (e.g., valvular disease) which as judged by the Investigator, may affect the patient's participation in or the outcome of this study.
* History of elective percutaneous coronary intervention (PCI) or coronary artery bypass grafting (CABG) within the past 6 months.
* History of clinically relevant or symptomatic cardiac arrhythmia such as sustained ventricular arrhythmia, non-fixed supra-ventricular arrhythmia which as judged by the Investigator, may affect the patient's participation in or the outcome of this study or which occurred within the past 6 months
* History of clinically relevant or symptomatic cardiac conduction abnormalities (any type of atrioventricular (AV) block, sick sinus syndrome, sinus node disease).
* Patients with a pacemaker or implantable cardioverter defibrillator.
* Known history of autoimmune disorders.
* Any severe viral, systemic, fungal, bacterial or protozoal infection within the past 6 months or chronic severe infection (hepatitis, HIV infection, tuberculosis).
* Presence of macular edema at fundus examination performed within 6 months before the first study drug administration.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2018-03-07 (Actual); Primary Completion 2018-12-22 (Actual); Study Completion 2018-12-22 (Actual)

PRIMARY OUTCOMES:
Change in Flow Mediated Dilation (FMD) | Baseline to Days 14, 21, 28, 35, and 42
  Absolute change from baseline in the % FMD index of the brachial artery

SECONDARY OUTCOMES:
Microvascular reactivity | Baseline to Days 14, 21, 28, 35, and 42
  Change from baseline in peak flow induced by acetylcholine iontophoresis measured using Laser Doppler perfusion monitoring
Number of adverse events | Up to Day 42
  Number of participants with adverse events
Assessment of pharmacokinetic (PK) parameter: Cmax | Days 1, 2, 3, 7, and 14
  Cmax: Maximum plasma concentration observed
Assessment of PK parameter: Ctrough | Days 1, 2, 3, 7, and 14
  Ctrough: Plasma concentration observed just before treatment administration during repeated dosing
Assessment of PK parameter: tmax | Days 1, 2, 3, 7, and 14
  tmax: Time to reach Cmax
Assessment of PK parameter: AUC0-24 | Days 1, 2, 3, 7, and 14
  AUC0-24: Area under the plasma concentration versus time curve over the dosing interval (24h)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (2):
- Germany (2):
  - Investigational Site Number 2760002, Mainz
  - Investigational Site Number 2760001, Neuss

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Bergougnan L, Andersen G, Plum-Morschel L, Evaristi MF, Poirier B, Tardat A, Ermer M, Herbrand T, Arrubla J, Coester HV, Sansone R, Heiss C, Vitse O, Hurbin F, Boiron R, Benain X, Radzik D, Janiak P, Muslin AJ, Hovsepian L, Kirkesseli S, Deutsch P, Parkar AA. Endothelial-protective effects of a G-protein-biased sphingosine-1 phosphate receptor-1 agonist, SAR247799, in type-2 diabetes rats and a randomized placebo-controlled patient trial. Br J Clin Pharmacol. 2021 May;87(5):2303-2320. doi: 10.1111/bcp.14632. Epub 2020 Nov 26. PMID 33125753